CLINICAL TRIAL: NCT00037752
Title: Use of Sibutramine in Smoking Cessation
Brief Title: Sibutramine to Reduce Weight Gain and Improve Smoking Cessation Rates
Acronym: SUCCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1176; R01HL068049 (NIH)
Record Dates: First submitted 2002-05-20; First posted 2002-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sibutramine plus a behavioral smoking cessation program
  Interventions: Drug: Sibutramine; Behavioral: Behavioral Smoking Cessation Program
- 2 (Active Comparator): Placebo sibutramine plus a behavioral smoking cessation program
  Interventions: Behavioral: Behavioral Smoking Cessation Program

INTERVENTIONS:
Drug: Sibutramine — At the baseline study visit, participants in Group 1 will be given a one month supply of 5 mg/d of sibutramine and a 1-month follow-up visit will be scheduled. After a safety evaluation at the 1-month follow-up visit, participants will have their dose of sibutramine titrated to 10 mg/d, a 1 month supply of the medication will be given to participants, and a 2-month follow-up visit will be scheduled. After a safety evaluation at the 2-month follow-up visit, participants will receive a 1 month supply of sibutramine 10 mg/d and a 3-month follow-up visit will be scheduled. At the 3-month follow-up visit, the sibutramine will be discontinued and participants will be scheduled for 4- and 5-month follow-up visits.
  Arms: 1
Behavioral: Behavioral Smoking Cessation Program — Both groups of participants will take part in a behavioral smoking cessation program.

SUMMARY:
The purpose of this study is to determine if sibutramine will decrease post-cessation weight gain and cigarette smoking in overweight and obese smokers who quit smoking.

DETAILED DESCRIPTION:
BACKGROUND:

Cigarette smoking poses a serious but preventable health risk. Behavioral smoking cessation programs have been shown to help individuals quit smoking. However, concerns about post-cessation weight gain have been reported as a significant barrier to quitting for many smokers. Recently, sibutramine, a new serotonin and norepinephrine reuptake inhibitor drug, has received FDA approval to help people lose weight. Since sibutramine affects neurotransmitters that are important in regulating body weight, it is reasonable to hypothesize that it may decrease post-cessation weight gain in overweight and obese smokers who quit smoking. To date, there have been no studies that compare sibutramine to a placebo, as a way to reduce post-cessation weight gain among overweight and obese smokers who take part in a behavioral smoking cessation program. Therefore, whether sibutramine is effective at reducing post-cessation weight gain in these smokers is unknown. Further, given the neuropharmacologic effects of sibutramine, it is reasonable to speculate that this medication could also be effective in helping individuals quit smoking both initially and in the long term. It is possible that the use of sibutramine, as compared to placebo, may result in a decrease in post-cessation weight gain in overweight and obese individuals who quit smoking. The use of sibutramine may also result in an increase in smoking cessation rates.

DESIGN NARRATIVE:

This study tests the hypothesis that the use of sibutramine, as compared to placebo, will result in a decrease in post-cessation weight gain in overweight and obese individuals who quit smoking, and result in an increase in smoking cessation rates. Participants will be randomly assigned to one of the following two groups: 1) sibutramine plus a behavioral smoking cessation program; or 2) placebo sibutramine plus a behavioral smoking cessation program. Assessments will include post-cessation weight change and smoking cessation rates measured during the study and 9 months following the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Body mass index greater than or equal to 25
* Currently smoke cigarettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2002-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Post-cessation weight change | Measured at 1 year follow-up
Smoking cessation | Measured at 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Karen C. Johnson, MD, MPH, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

REFERENCES:
- [Result] DeBon M, Johnson KC, Bush A, and Klesges RC. (2008, March). The efficacy of sibutramine to prevent or decrease post cessation weight gain in overweight and obese smokers. Paper presented at the 29th annual meeting of the Society of Behavioral Medicine, San Diego, CA. March 2008.